CLINICAL TRIAL: NCT02239679
Title: A Phase 2 Study Comparing the Occurrence of Actinic Keratoses on the Face in High-Risk Individuals After Cryotherapy + Photodynamic Therapy With Levulan Topical Solution + Blue Light Versus Cryotherapy + Vehicle Topical Solution + Blue Light
Brief Title: Controlled Study of the Occurrence of Actinic Keratosis on the Face After Cryotherapy + Aminolevulinic Acid (ALA) Photodynamic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP0109
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2017-09

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Solutions; Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALA X3 (Experimental): Cryotherapy followed by 3 aminolevulinic acid + blue light (BLU-U) treatments
  Interventions: Drug: Aminolevulinic Acid; Device: BLU-U; Procedure: Cryotherapy
- VEH (Placebo Comparator): Vehicle (VEH) group will be randomized (1:1) to be balanced for the two active groups; receiving cryotherapy and 2 or 3 subsequent Topical Solution Vehicle + BLU-U treatments. Subjects receiving VEH will be considered a single treatment group.
  Interventions: Drug: Topical Solution Vehicle; Device: BLU-U; Procedure: Cryotherapy
- ALA X2 (Experimental): Cryotherapy followed by 2 aminolevulinic acid + BLU-U treatments
  Interventions: Drug: Aminolevulinic Acid; Device: BLU-U; Procedure: Cryotherapy

INTERVENTIONS:
Drug: Aminolevulinic Acid — 20% ALA applied to face for one hour prior to 10 J/cm2 blue light
  Other Names: Levulan Kerastick; ALA
  Arms: ALA X2; ALA X3
Drug: Topical Solution Vehicle — Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to face one hour prior to 10 J/cm2 blue light
  Arms: VEH
Device: BLU-U — 10 J/cm2 blue light delivered at 10 mW/cm2
  Other Names: BLU-U Blue Light Photodynamic Therapy Illuminator
Procedure: Cryotherapy — Liquid nitrogen cryotherapy by standard of care method to all visible/palpable actinic keratosis (AK) lesions at screening.
  Other Names: Liquid Nitrogen

SUMMARY:
The purpose of this study is to determine if Levulan photodynamic therapy (PDT) is safe and effective in the treatment of actinic keratoses (AK) on the face, following treatment with liquid nitrogen cryotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Four to fifteen AKs on the face
* histologically confirmed presence of abnormal architecture and satellite atypical keratinocytes in the epidermis, in clinically normal tissue samples of photodamaged skin adjacent to AKs
* at least one previously treated nonmelanoma skin cancer (NMSC) on the head and/or neck area within the past five years

Exclusion Criteria:

* Pregnancy
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the Treatment Area
* skin pathology or condition which could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy
* Subject is immunosuppressed
* unsuccessful outcome from previous ALA-PDT therapy
* currently enrolled in an investigational drug or device study
* has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment
* known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol)
* has an active herpes simplex infection OR a history of 2 or more outbreaks within the past 12 months, on the face
* use of the following topical preparations on the extremity to be treated:

  * Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g.glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days
  * Retinoids, including tazarotene, adapalene, tretinoin, within 4 weeks
  * Microdermabrasion, laser ablative treatments, ALA-PDT, chemical peels, 5-fluorouracil (5-FU), diclofenac, ingenol mebutate, imiquimod or other topical treatments for AK within 8 weeks
* use of systemic retinoid therapy within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, MD, PhD, Study Director — DUSA Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - UCSD Dermatology, San Diego, California
  - Therapeutics Clinical Research, San Diego, California
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Shideler Clinical Research Center, Carmel, Indiana
  - Sadick Research Group, New York, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Suzanne Bruce and Associates, P.A.,The Center for Skin Research, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- [Derived] Piacquadio D, Berman B, Siegel DM, Bhatia N, Brocato J, Squittieri N, Pariser DM. Treatment Satisfaction and Acceptability of 20% Aminolevulinic Acid Photodynamic Therapy for the Treatment of Actinic Keratoses of the Face, Scalp, and Upper Extremities. J Clin Aesthet Dermatol. 2023 Dec;16(12):46-51. PMID 38125671

RESULTS

PARTICIPANT FLOW:
Groups:
- ALA X2: Cryotherapy followed by 2 aminolevulinic acid + blue light (BLU-U) treatments
  Aminolevulinic Acid: 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  BLU-U: 10 J/cm2 blue light delivered at 10 mW/cm2
  Cryotherapy: Liquid nitrogen cryotherapy by standard of care method to all visible/palpable actinic keratosis (AK) lesions at screening.
- ALA X3: Cryotherapy followed by 3 aminolevulinic acid + BLU-U treatments
  Aminolevulinic Acid: 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  BLU-U: 10 J/cm2 blue light delivered at 10 mW/cm2
  Cryotherapy: Liquid nitrogen cryotherapy by standard of care method to all visible/palpable AK lesions at screening.
- VEH-PDT: Vehicle (VEH) group will be randomized (1:1) to be balanced for the two active groups; receiving cryotherapy and 2 or 3 subsequent Topical Solution Vehicle + BLU-U treatments. Subjects receiving VEH will be considered a single treatment group.
  Topical Solution Vehicle: Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to upper extremities 3 hours prior to 10 J/cm2 blue light
  BLU-U: 10 J/cm2 blue light delivered at 10 mW/cm2
  Cryotherapy: Liquid nitrogen cryotherapy by standard of care method to all visible/palpable AK lesions at screening.
Period: Overall Study
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Started | 53 | 59 | 54
Completed | 50 | 56 | 53
Not Completed | 3 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- ALA X2: Cryotherapy followed by 2 aminolevulinic acid + BLU-U treatments
  Aminolevulinic Acid: 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  BLU-U: 10 J/cm2 blue light delivered at 10mW/cm2
  Cryotherapy: Liquid nitrogen cryotherapy by standard of care method to all visible/palpable AK lesions at screening.
- ALA X3: Cryotherapy followed by 3 aminolevulinic acid + BLU-U treatments
  Aminolevulinic Acid: 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  BLU-U: 10 J/cm2 blue light delivered at 10mW/cm2
  Cryotherapy: Liquid nitrogen cryotherapy by standard of care method to all visible/palpable AK lesions at screening.
- VEH-PDT: Vehicle (VEH) group will be randomized (1:1) to be balanced for the two active groups; receiving cryotherapy and 2 or 3 subsequent Topical Solution Vehicle + BLU-U treatments. Subjects receiving VEH will be considered a single treatment group.
  Topical Solution Vehicle: Levulan Kerastick containing vehicle ingredients only. Vehicle solution applied to upper extremities 3 hours prior to 10 J/cm2 blue light
  BLU-U: 10 J/cm2 blue light delivered at 10mW/cm2
  Cryotherapy: Liquid nitrogen cryotherapy by standard of care method to all visible/palpable AK lesions at screening.
- Total: Total of all reporting groups
Arm/Group | ALA X2 | ALA X3 | VEH-PDT | Total
Number analyzed (Participants) | 53 | 59 | 54 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.65) | 66.7 (9.35) | 65.8 (9.5) | 66.8 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 10 | 31
  Male | 43 | 48 | 44 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 52 | 59 | 53 | 164
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 53 | 59 | 54 | 166
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 59 | 54 | 166
Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type staging:
  Skin Type I - Burns easily, never tans Skin Type II - Burns easily, tans minimally Skin Type III - Burns moderately, tans gradually Skin Type IV - Burns minimally, tans well Skin Type V - Rarely burns, tans profusely
  Participants
    Skin Type I - Burns easily, never tans | 6 | 5 | 2 | 13
    Skin Type II - Burns easily, tans minimally | 29 | 37 | 35 | 101
    Skin Type III - Burns moderately, tans gradually | 16 | 12 | 12 | 40
    Skin Type IV - Burns minimally, tans well | 2 | 4 | 5 | 11
    Skin Type V - Rarely burns, tans profusely | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Number of AKs in Treatment Area
Description: Count of observed lesions in the treatment area, which include lesions that recurred after on-study cryotherapy as well as newly occurring lesions. AK lesions in the treatment area at baseline (maximum of 2) were excluded for this endpoint.
Time Frame: Week 52
Population: Analysis population consisted of observed data; ie. subjects remaining on-study at Week 52.
Measure: Least Squares Mean (Standard Error); unit: lesions
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
lesions | 3.0 (0.91) | 2.1 (0.84) | 4.7 (0.86)
Statistical Analysis 1: Comparison: ALA X3 vs VEH-PDT; Test type: Superiority; p = 0.0166, ANCOVA

2. Secondary Outcome: Proportion of Subjects With 0 AKs
Description: Normalized based on number of lesions present at Baseline
Time Frame: Week 4
Population: Analysis population consisted of observed data; ie. subjects with data at Week 4.
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 54
Participants | 35 | 35 | 27

3. Secondary Outcome: Subject Satisfaction Score
Description: Subject satisfaction score
  1. = Excellent (very satisfied)
  2. = Good (moderately satisfied)
  3. = Fair (slightly satisfied)
  4. = Poor (not satisfied at all) Unknown
Time Frame: Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Very Satisfied | 27 | 26 | 16
  Moderately Satisfied | 15 | 21 | 14
  Slightly Satisfied | 7 | 9 | 14
  Not Satisfied | 2 | 0 | 9
  Unknown | 2 | 3 | 1

4. Secondary Outcome: Proportion of Subjects With 0 AKs
Description: Normalized based on number of lesions present at Baseline
Time Frame: Week 12
Population: Analysis population consisted of observed data; ie. subjects with data at Week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 53
Participants | 27 | 35 | 22

5. Secondary Outcome: Proportion of Subjects With 0 AKs
Description: Normalized based on number of lesions present at Baseline
Time Frame: Week 24
Population: Analysis population consisted of observed data only.
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 56 | 53
Participants | 30 | 22 | 14

6. Secondary Outcome: Proportion of Subjects With 0 AKs
Description: Normalized based on number of lesions present at Baseline
Time Frame: Week 36
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants | 15 | 20 | 10

7. Secondary Outcome: Proportion of Subjects With 0 AKs
Description: Normalized based on number of lesions present at Baseline
Time Frame: Week 52
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants | 18 | 21 | 10
Statistical Analysis 1: Comparison: ALA X2 vs VEH-PDT; Test type: Superiority; p = 0.0102, Cochran-Mantel-Haenszel — no adjustments for multiple comparisons; stratified by site
Statistical Analysis 2: Comparison: ALA X3 vs VEH-PDT; Test type: Superiority; p = 0.0089, Cochran-Mantel-Haenszel — no adjustment for multiple comparisons; stratified by site

8. Secondary Outcome: Recurrence Rate
Description: Recurrence rate of all lesions that were complete responses following on-study cryotherapy (at Visit 3/Baseline).
Time Frame: Week 52
Population: Analysis population consisted of observed data only
Measure: Count of Units; unit: number of lesions
Units Other Than Participants: number of lesions
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Number analyzed (number of lesions) | 441 | 525 | 522
number of lesions | 34 | 32 | 81
Statistical Analysis 1: Comparison: ALA X2 vs VEH-PDT; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — no adjustments for multiple comparisons; stratified by site
Statistical Analysis 2: Comparison: ALA X3 vs VEH-PDT; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — no adjustment for multiple comparison; stratified by site

9. Secondary Outcome: Duration of Response
Description: Duration of response is the elapsed number of weeks from the Baseline visit until a lesion recurred or Week 52, whichever comes first
Time Frame: within 52 weeks after Baseline
Population: Subjects who discontinued prior to Week 52 were excluded; analysis used observed data only.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
weeks | 35.9 (20.4) | 33.3 (19.7) | 25.9 (20.7)

10. Other Pre Specified Outcome: Hyperpigmentation
Description: HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Time Frame: Screening
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 22 | 27 | 25
  Grade 1 | 17 | 23 | 20
  Grade 2 | 13 | 5 | 8
  Grade 3 | 1 | 3 | 1
  Grade 4 | 0 | 1 | 0

11. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 23 | 26 | 22
  Grade 1 | 17 | 25 | 22
  Grade 2 | 12 | 5 | 9
  Grade 3 | 1 | 2 | 1
  Grade 4 | 0 | 1 | 0

12. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: 24-48 hours after photodynamic therapy (PDT) #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 57 | 53
Participants
  Grade 0 | 23 | 22 | 23
  Grade 1 | 14 | 24 | 21
  Grade 2 | 13 | 10 | 8
  Grade 3 | 3 | 0 | 1
  Grade 4 | 0 | 1 | 0

13. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: 4 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 54
Participants
  Grade 0 | 21 | 26 | 23
  Grade 1 | 21 | 25 | 23
  Grade 2 | 8 | 4 | 7
  Grade 3 | 1 | 1 | 1
  Grade 4 | 0 | 1 | 0

14. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: 12 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 53
Participants
  Grade 0 | 22 | 28 | 23
  Grade 1 | 21 | 22 | 23
  Grade 2 | 8 | 5 | 6
  Grade 3 | 0 | 1 | 1
  Grade 4 | 0 | 1 | 0

15. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: 24 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 56 | 53
Participants
  Grade 0 | 25 | 26 | 24
  Grade 1 | 18 | 24 | 23
  Grade 2 | 8 | 4 | 5
  Grade 3 | 0 | 1 | 1
  Grade 4 | 0 | 1 | 0

16. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: 36 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 24 | 25 | 24
  Grade 1 | 19 | 26 | 23
  Grade 2 | 7 | 3 | 5
  Grade 3 | 0 | 1 | 1
  Grade 4 | 0 | 1 | 0

17. Other Pre Specified Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: 52 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 22 | 24 | 24
  Grade 1 | 21 | 25 | 23
  Grade 2 | 7 | 5 | 5
  Grade 3 | 0 | 1 | 1
  Grade 4 | 0 | 1 | 0

18. Other Pre Specified Outcome: Hypopigmentation
Description: HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation
Time Frame: Screening
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 35 | 40 | 38
  Grade 1 | 16 | 17 | 14
  Grade 2 | 2 | 2 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

19. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 18
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 37 | 38 | 37
  Grade 1 | 14 | 19 | 14
  Grade 2 | 2 | 2 | 3
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

20. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 18
Time Frame: 24-48 hours after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 57 | 53
Participants
  Grade 0 | 34 | 35 | 35
  Grade 1 | 14 | 19 | 16
  Grade 2 | 4 | 2 | 2
  Grade 3 | 1 | 1 | 0
  Grade 4 | 0 | 0 | 0

21. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 18
Time Frame: 4 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 54
Participants
  Grade 0 | 34 | 38 | 35
  Grade 1 | 14 | 17 | 17
  Grade 2 | 3 | 2 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

22. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 18
Time Frame: 12 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 53
Participants
  Grade 0 | 33 | 40 | 35
  Grade 1 | 14 | 15 | 17
  Grade 2 | 4 | 1 | 1
  Grade 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0

23. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 18
Time Frame: 24 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 56 | 53
Participants
  Grade 0 | 33 | 39 | 37
  Grade 1 | 16 | 15 | 15
  Grade 2 | 2 | 1 | 1
  Grade 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0

24. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 18
Time Frame: 36 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 31 | 38 | 35
  Grade 1 | 18 | 16 | 17
  Grade 2 | 1 | 1 | 1
  Grade 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0

25. Other Pre Specified Outcome: Hypopigmentation
Description: as for outcome 18
Time Frame: 52 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 26 | 35 | 33
  Grade 1 | 22 | 19 | 19
  Grade 2 | 2 | 1 | 1
  Grade 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0

26. Other Pre Specified Outcome: Erythema
Description: Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Screening
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 31 | 41 | 33
  Grade 1 | 16 | 13 | 13
  Grade 2 | 6 | 4 | 8
  Grade 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0

27. Other Pre Specified Outcome: Erythema
Description: as for outcome 26
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 34 | 38 | 33
  Grade 1 | 14 | 18 | 15
  Grade 2 | 5 | 3 | 6
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

28. Other Pre Specified Outcome: Erythema
Description: as for outcome 26
Time Frame: 5 minutes after PDT #1
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 4 | 6 | 11
  Grade 1 | 8 | 11 | 27
  Grade 2 | 29 | 25 | 12
  Grade 3 | 12 | 17 | 4
  Grade 4 | 0 | 0 | 0

29. Other Pre Specified Outcome: Erythema
Description: as for outcome 26
Time Frame: 24-48 hours after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 57 | 53
Participants
  Grade 0 | 2 | 3 | 22
  Grade 1 | 12 | 10 | 21
  Grade 2 | 13 | 14 | 8
  Grade 3 | 23 | 26 | 2
  Grade 4 | 3 | 4 | 0

30. Other Pre Specified Outcome: Erythema
Description: as for outcome 26
Time Frame: 4 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 54
Participants
  Grade 0 | 35 | 41 | 34
  Grade 1 | 14 | 14 | 15
  Grade 2 | 2 | 2 | 5
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

31. Other Pre Specified Outcome: Erythema
Description: as for outcome 26
Time Frame: 12 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 53
Participants
  Grade 0 | 35 | 43 | 36
  Grade 1 | 16 | 13 | 15
  Grade 2 | 0 | 1 | 1
  Grade 3 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0

32. Other Pre Specified Outcome: Erythema
Description: as for outcome 26
Time Frame: 24 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 56 | 53
Participants
  Grade 0 | 37 | 41 | 31
  Grade 1 | 14 | 13 | 20
  Grade 2 | 0 | 2 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

33. Other Pre Specified Outcome: Erythema
Description: as for outcome 26
Time Frame: 36 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 37 | 36 | 33
  Grade 1 | 13 | 19 | 18
  Grade 2 | 0 | 1 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

34. Other Pre Specified Outcome: Erythema
Description: as for outcome 26
Time Frame: 52 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 38 | 40 | 37
  Grade 1 | 11 | 14 | 14
  Grade 2 | 1 | 2 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

35. Other Pre Specified Outcome: Edema
Description: EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Time Frame: Screening
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 52 | 59 | 54
  Grade 1 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

36. Other Pre Specified Outcome: Edema
Description: as for outcome 35
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 53 | 59 | 54
  Grade 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

37. Other Pre Specified Outcome: Edema
Description: as for outcome 35
Time Frame: 5 minutes after PDT #1
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 46 | 44 | 52
  Grade 1 | 6 | 12 | 2
  Grade 2 | 1 | 2 | 0
  Grade 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0

38. Other Pre Specified Outcome: Edema
Description: as for outcome 35
Time Frame: 24-48 hours after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 57 | 53
Participants
  Grade 0 | 33 | 31 | 53
  Grade 1 | 14 | 16 | 0
  Grade 2 | 6 | 10 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

39. Other Pre Specified Outcome: Edema
Description: as for outcome 35
Time Frame: 4 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 54
Participants
  Grade 0 | 51 | 56 | 53
  Grade 1 | 0 | 0 | 1
  Grade 2 | 0 | 1 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

40. Other Pre Specified Outcome: Edema
Description: as for outcome 35
Time Frame: 12 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 53
Participants
  Grade 0 | 51 | 57 | 53
  Grade 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

41. Other Pre Specified Outcome: Edema
Description: as for outcome 35
Time Frame: 24 weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 56 | 53
Participants
  Grade 0 | 51 | 56 | 53
  Grade 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

42. Other Pre Specified Outcome: Edema
Description: as for outcome 35
Time Frame: 36 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 49 | 55 | 51
  Grade 1 | 1 | 1 | 1
  Grade 2 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

43. Other Pre Specified Outcome: Edema
Description: as for outcome 35
Time Frame: 52 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 50 | 56 | 53
  Grade 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

44. Other Pre Specified Outcome: Stinging/Burning
Description: STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: Screening
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 53 | 58 | 53
  Grade 1 | 0 | 1 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

45. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 44
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 53 | 59 | 53
  Grade 1 | 0 | 0 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

46. Other Pre Specified Outcome: Stinging/Burning
Description: Immediately after PDT, the most intensive, acute perception of Stinging/Burning DURING treatment will be recorded.
  STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: During PDT #1
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 5 | 5 | 42
  Grade 1 | 18 | 21 | 11
  Grade 2 | 27 | 32 | 1
  Grade 3 | 3 | 1 | 0

47. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 44
Time Frame: 5 minutes after PDT #1
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 11 | 11 | 46
  Grade 1 | 33 | 37 | 8
  Grade 2 | 9 | 11 | 0
  Grade 3 | 0 | 0 | 0

48. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 44
Time Frame: 24-48 hours after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 57 | 53
Participants
  Grade 0 | 31 | 23 | 51
  Grade 1 | 17 | 29 | 2
  Grade 2 | 5 | 5 | 0
  Grade 3 | 0 | 0 | 0

49. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 44
Time Frame: 4 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 54
Participants
  Grade 0 | 51 | 57 | 53
  Grade 1 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0

50. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 44
Time Frame: 12 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 53
Participants
  Grade 0 | 51 | 57 | 52
  Grade 1 | 0 | 0 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0

51. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 44
Time Frame: 24 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 56 | 53
Participants
  Grade 0 | 51 | 55 | 53
  Grade 1 | 0 | 1 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0

52. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 44
Time Frame: 36 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 49 | 56 | 51
  Grade 1 | 0 | 0 | 2
  Grade 2 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0

53. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 44
Time Frame: 52 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 49 | 56 | 52
  Grade 1 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0

54. Other Pre Specified Outcome: Scaling & Dryness
Description: SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Time Frame: Screening
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 41 | 43 | 40
  Grade 1 | 8 | 11 | 11
  Grade 2 | 4 | 4 | 3
  Grade 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0

55. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 54
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 38 | 44 | 39
  Grade 1 | 10 | 12 | 11
  Grade 2 | 4 | 3 | 4
  Grade 3 | 1 | 0 | 0
  Grade 4 | 0 | 0 | 0

56. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 54
Time Frame: 24-48 hours after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 57 | 53
Participants
  Grade 0 | 30 | 35 | 38
  Grade 1 | 18 | 14 | 13
  Grade 2 | 4 | 7 | 2
  Grade 3 | 1 | 1 | 0
  Grade 4 | 0 | 0 | 0

57. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 54
Time Frame: 4 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 54
Participants
  Grade 0 | 41 | 46 | 41
  Grade 1 | 10 | 10 | 11
  Grade 2 | 0 | 1 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

58. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 54
Time Frame: 12 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 53
Participants
  Grade 0 | 40 | 44 | 43
  Grade 1 | 10 | 11 | 7
  Grade 2 | 0 | 2 | 2
  Grade 3 | 1 | 0 | 1
  Grade 4 | 0 | 0 | 0

59. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 54
Time Frame: 24 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 56 | 53
Participants
  Grade 0 | 43 | 46 | 39
  Grade 1 | 6 | 8 | 12
  Grade 2 | 2 | 2 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

60. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 54
Time Frame: 36 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 38 | 46 | 38
  Grade 1 | 11 | 8 | 13
  Grade 2 | 1 | 2 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

61. Other Pre Specified Outcome: Scaling & Dryness
Description: as for outcome 54
Time Frame: 52 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 42 | 42 | 47
  Grade 1 | 6 | 10 | 4
  Grade 2 | 2 | 4 | 2
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

62. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Time Frame: Screening
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 53 | 58 | 53
  Grade 1 | 0 | 1 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

63. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 62
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 59 | 54
Participants
  Grade 0 | 49 | 58 | 51
  Grade 1 | 4 | 1 | 2
  Grade 2 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

64. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 62
Time Frame: 24-48 hours after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 53 | 57 | 53
Participants
  Grade 0 | 50 | 53 | 49
  Grade 1 | 3 | 3 | 3
  Grade 2 | 0 | 0 | 1
  Grade 3 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0

65. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 62
Time Frame: 4 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 54
Participants
  Grade 0 | 51 | 56 | 51
  Grade 1 | 0 | 1 | 2
  Grade 2 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

66. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 62
Time Frame: 12 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 57 | 53
Participants
  Grade 0 | 50 | 56 | 53
  Grade 1 | 1 | 1 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

67. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 62
Time Frame: 24 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 51 | 56 | 53
Participants
  Grade 0 | 50 | 56 | 53
  Grade 1 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

68. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 62
Time Frame: 36 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 50 | 56 | 52
  Grade 1 | 0 | 0 | 1
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

69. Other Pre Specified Outcome: Oozing/Vesiculation/Crusting
Description: as for outcome 62
Time Frame: 52 Weeks after PDT #1
Population: Analysis population consisted of observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
Number analyzed (Participants) | 50 | 56 | 53
Participants
  Grade 0 | 49 | 56 | 53
  Grade 1 | 1 | 0 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | ALA X2 | ALA X3 | VEH-PDT
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/59 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/53 | 3/59 | 4/54
Other Adverse Events (participants affected / at risk) | 13/53 | 9/59 | 15/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALA X2 (N=53) | ALA X3 (N=59) | VEH-PDT (N=54)
acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
angina unstable (Cardiac disorders) | 0 | 1 | 0
atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
coronary artery disease (Cardiac disorders) | 0 | 0 | 1
vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
headache (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALA X2 (N=53) | ALA X3 (N=59) | VEH-PDT (N=54)
procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 3
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 5 | 4
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of results will be made by the Sponsor. If publication is not submitted within 12 months after the date of study final report, the PI may publish the results from the site individually, subject to compliance with the other terms of the clinical trial agreement, including a requirement that the PI provide a draft of the publication for the sponsor's review 30 days before submission for publication so that sponsor can review the publication for confidential information